CLINICAL TRIAL: NCT07283120
Title: The Impact of Breast Surgery on Patients' Quality of Life
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00210; bb25kappos3
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to document the surgery-specific and overall Quality of life parameters of patients undergoing all types of breast surgery at the University Hospital of Basel

DETAILED DESCRIPTION:
The planned ten-year follow-up using Patient reported outcome measure will give us the unique opportunity to gain insight into patients' breast-related QoL (Quality of Life) long after surgery and detect systematic issues that may affect them beyond the scope of routine follow-up consultations. Along with the detection of any occurring adverse events, the information gathered in the database will facilitate the search for risk factors involved in their development, ideally resulting in their rectification and thus contributing to patient well-being in the long term.

ELIGIBILITY:
Inclusion Criteria:

* adults who underwent any type of breast surgery at the University Hospital of Basel

Exclusion Criteria:

* Patients under the age of 18 years, without general consent or written informed consent, with insufficient language comprehension or other factors limiting their ability to co-operate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent breast surgery at the University Hospital Basel from 2014 onwards
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2035-06-30 (Estimated); Study Completion 2035-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | up to 10 years
  five point likert-scale for satisfaction ( psychometric survey response scale ranging from "Strongly Disagree" to "Strongly Agree". The format includes: 1. Strongly Disagree, 2. Disagree, 3. Neutral (or Neither Agree nor Disagree), 4. Agree, and 5. Strongly Agree Descriptive measures using patient-reported outcome measures (BREAST-Q, McGill short form, EQ-5D-5L)
Patient reported quality of life | up to 10 years
  Descriptive measures using patient-reported outcome measures (BREAST-Q, McGill short form, EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kappos, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland